CLINICAL TRIAL: NCT03735069
Title: Outcome of Vital Pulp Therapy in Carious Teeth With Hypomineralization Defects: a Clinical Study
Brief Title: Vital Pulp Therapy in Carious Teeth With Hypomineralization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Ola B. Al-Batayneh, Associate Professor, Jordan University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 77-2017
Record Dates: First submitted 2018-11-04; First posted 2018-11-08 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Dental Caries Extending to Pulp; Molar Incisor Hypomineralization
Keywords: Vital pulp therapy; Indirect pulp treatment; Partial (Cvek) pulpotomy; Complete (cervical) pulpotomy; Enamel hypomineralization defects; Molar incisor hypomineralization; Children
MeSH Terms: conditions — Molar Hypomineralization | interventions — adenylate isopentenyltransferase

STUDY DESIGN:
Intervention Model Description: The study will be a prospective case series study; VPT (IPT, partial or complete pulpotomies) will be done depending on the severity of the case (depth of caries/pulpal involvement, symptoms and response to vitality testing). The study will include about 150 hypomineralized first permanent molars, patients age will range from 6-16 years old. Sample will be divided into 3 groups according to the treatment that will be provided (IPT / Cvek pulpotomy / Cervical pulpotomy). Patients' teeth will be randomly allocated to different treatment procedures (IPT or pulpotomy) using random tables.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- IPT (Indirect pulp treatment) group (Experimental): In this group, complete caries excavation from the dentin-enamel junction will be done. Caries near the pulp will be removed with caution until the remaining dentin shows increased resistance to manual instrumentation. A layer of resin-modified glass ionomer (RMGI) dressing material will be placed (Vitrebond; St.Paul, MN), followed by resin-modified glass ionomer (RMGI) build-up material (Vitremer; St. Paul, MN), and the final restoration of choice for MIH involved teeth; a preformed Stainless Steel Crown (SSC).
  Interventions: Procedure: IPT (Indirect pulp treatment)
- Cvek/partial pulpotomy group (Experimental): In this group, partial pulpotomy will be attempted first, inflamed pulp tissue will be removed until healthy pulp tissue is reached (2-4mm depth), as indicated by healthy bleeding and arrest of hemorrhage upon pressure with a cotton pellet moistened with 2.5% NaOCl for 2-5 minutes and repeated twice if required; otherwise, cervical pulpotomy will be done.
  Gray MTA (Mineral Trioxide Aggregate, Dentsply, Canada) will be placed in the pulp chamber (2-3mm thickness), a moist cotton pellet will be placed and Intermediate Restorative Material (IRM) to ensure setting. Patient will be reviewed after 1 week. If the tooth is asymptomatic, final restoration with RMGI (Vitremer; St. Paul, MN) and stainless steel crown will be placed , and a post-op radiograph will be taken.
  Interventions: Procedure: Cvek/partial pulpotomy
- Cervical pulpotomy group (Experimental): In this group, a cervical pulpotomy procedure will be done where all pulp chamber tissue shall be removed until healthy pulp tissue is reached, as indicated by bleeding from all canals and arrest of hemorrhage upon pressure (for maximum 6 minutes).
  Gray MTA (Mineral Trioxide Aggregate, Dentsply, Canada) will be mixed according to manufacturer instructions and will be placed in the pulp chamber in 2-3 mm thickness, moist cotton pellet will be placed to ensure setting and the tooth will be temporized with Intermediate Restorative Material (IRM), the patient will be reviewed after 1 week. If the tooth is asymptomatic, final restoration with RMGI (Vitremer; St. Paul, MN) and stainless steel crown will be placed , and a post-op radiograph will be taken.
  Interventions: Procedure: Cervical pulpotomy

INTERVENTIONS:
Procedure: IPT (Indirect pulp treatment) — Indirect pulp treatment involves complete caries excavation from the dentin-enamel junction using a round bur. Caries near the pulp is removed with caution using spoon excavator until the remaining dentine shows increased resistance to manual instrumentation. A layer of resin-modified glass ionomer (RMGI) dressing material is placed, followed by resin-modified glass ionomer (RMGI) build-up material, and the final restoration; a preformed Stainless Steel Crown (SSC).
  Other Names: Indirect pulp capping
  Arms: IPT (Indirect pulp treatment) group
Procedure: Cvek/partial pulpotomy — Cvek/partial pulpotomy involves removal of inflamed pulp tissue to depth until healthy pulp tissue is reached (depth of 2-4 mm), as indicated by healthy bleeding and arrest of hemorrhage upon pressure with a cotton pellet moistened with 2.5% NaOCl for 2-5 minutes and repeated for two times if required. Gray MTA will be placed in the pulp chamber in 2-3 mm thickness, moist cotton pellet will be placed to ensure setting and the tooth will be temporized with IRM, the patient will be reviewed after 1 week. If the tooth is asymptomatic, final restoration with RMGIC and stainless steel crown will be placed , and a post-operative radiograph will be taken.
  Arms: Cvek/partial pulpotomy group
Procedure: Cervical pulpotomy — Cervical pulpotomy involves removal of inflamed pulp tissue from all pulp chamber as indicated by healthy bleeding and arrest of hemorrhage upon pressure with a cotton pellet moistened with 2.5% NaOCl for 6 minutes and repeated for two times if required. Gray MTA will be placed in the pulp chamber (2-3mm) thickness, moist cotton pellet will be placed to ensure setting and the tooth will be temporized with IRM, the patient will be reviewed after 1 week. If the tooth is asymptomatic, final restoration with RMGIC and stainless steel crown will be placed , and a post-operative radiograph will be taken.
  Arms: Cervical pulpotomy group

SUMMARY:
Vital pulp therapy (VPT) is a general term for multiple procedures (indirect pulp cap, direct pulp cap and pulpotomy) all directed toward preserving pulp vitality and enable complete root development in immature teeth. The aim of this study is to evaluate the clinical, radiographic and histologic (if any teeth later are doomed for extraction for orthodontic or other reasons) success rate of VPT on treating cariously exposed permanent teeth with developmental defects of enamel. This will be a a prospective case series study including children between 6-16 years old having tooth with enamel hypomineralization defect with deep caries, restorable teeth , and no signs of infection. The teeth will be followed up both clinically and radiographically for 1 year after treatment. It is expected that the teeth will maintain vitality with resolution of symptoms (if present) and completion of root development in immature teeth after vital pulp therapy.

DETAILED DESCRIPTION:
Background: One of the greatest challenges that may affect the integrity of teeth is dental caries. If left untreated, pulpal involvement may occur leading to irreversible damage and eventually necrosis. This risk is greatly increased in the presence of developmental defects affecting tooth enamel such as molar-incisor hypomineralization (MIH). Despite having high success rate, root canal treatment will lead to loss of proprioceptive function, loss of stress-reducing damping property and tooth sensitivity in developed teeth and will also inhibit complete root formation in immature permanent teeth. Vital pulp therapy (VPT) is a general term for multiple procedures (indirect pulp cap, direct pulp cap and pulpotomy) all directed toward preserving pulp vitality and enable complete root development in immature teeth. So, it has been advocated as a better alternative for pulpectomy/root canal treatment in deep carious vital permanent teeth.

Aim: To evaluate the clinical, radiographic and histologic (if any teeth later are doomed for extraction for orthodontic or other reasons) success rate of VPT on treating cariously exposed permanent teeth with developmental defects of enamel.

Materials and methods: The study will be a prospective case series study including children between 6-16 years old. Inclusion criteria include patients having tooth with enamel hypomineralization defect with deep caries. Teeth should be restorable tooth. No soft tissue swellings, mobility or tenderness to percussion should be present. In cases of pulpotomy, bleeding from all canals should be present after opening the access. Tooth should be diagnosed with reversible / irreversible pulpitis (as indicated by positive response to cold testing).

Medically compromised patients will be excluded from the study. Also any tooth that is non-restorable, having sinus tract or periodontally compromised will be excluded. The procedure involves taking preoperative compete records (radiograph, vitality tests, percussion, mobility and photographs). After administration of anesthetic agent, rubber dam will be placed, caries is removed and appropriate dressing pulp material will be placed and then the final restoration is placed. A post-operative x-ray will be taken. The teeth will be followed up both clinically and radiographically for 1 year after treatment.

Expected Results: It is expected that the teeth will maintain vitality with resolution of symptoms (if present) and completion of root development in immature teeth after vital pulp therapy.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patient between 6-16 years.
* Tooth with enamel hypomineralization defect
* Molar tooth with deep caries
* Restorable molar tooth
* No soft tissue swellings, mobility or tenderness to percussion
* Bleeding from all canals (when performing cervical pulpotomy)
* Reversible / Irreversible pulpitis (as indicated by positive response to pulp testing using cold test)

Exclusion Criteria:

* Medically compromised patient
* Non-restorable tooth
* Presence of dental abcess / sinus tract
* Periodontally compromised teeth

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Clinical Success | 12 months
  Clinical parameters indicating successful treatment include the following criteria:
  * Absence of symptoms (except on the first 24 hrs)
  * No tenderness to percussion
  * Normal soft tissue around the tooth (no swellings or sinus tract)
  * Reduction in PAI if rarefaction was present
  * Normal response to cold test
  * Continued root development (immature teeth)
Radiographic Success | 12 months
  Radiographic parameters indicating successful treatment is based on the periapical index (PAI), and includes 5 scores from 1-5:
  PAI 1 - normal periapical structure PAI 2 - small changes in bone structure not pathognomic for apical periodontitis PAI 3 - changes in bone structure with some mineral loss characteristic of apical periodontitis PAI 4 - periodontitis with well defined radiolucent area PAI 5 - severe periodontitis with exacerbating features and bone expansion

CONTACTS AND LOCATIONS:
Overall Officials: Ola Al-Batayneh, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- Jordan University of Science and Technology, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aguilar P, Linsuwanont P. Vital pulp therapy in vital permanent teeth with cariously exposed pulp: a systematic review. J Endod. 2011 May;37(5):581-7. doi: 10.1016/j.joen.2010.12.004. Epub 2011 Mar 5. PMID 21496652
- [Background] Asgary S, Shahabi S, Jafarzadeh T, Amini S, Kheirieh S. The properties of a new endodontic material. J Endod. 2008 Aug;34(8):990-3. doi: 10.1016/j.joen.2008.05.006. Epub 2008 Jun 20. PMID 18634932
- [Background] Bjorndal L, Reit C, Bruun G, Markvart M, Kjaeldgaard M, Nasman P, Thordrup M, Dige I, Nyvad B, Fransson H, Lager A, Ericson D, Petersson K, Olsson J, Santimano EM, Wennstrom A, Winkel P, Gluud C. Treatment of deep caries lesions in adults: randomized clinical trials comparing stepwise vs. direct complete excavation, and direct pulp capping vs. partial pulpotomy. Eur J Oral Sci. 2010 Jun;118(3):290-7. doi: 10.1111/j.1600-0722.2010.00731.x. PMID 20572864
- [Background] Farsi N, Alamoudi N, Balto K, Al Mushayt A. Clinical assessment of mineral trioxide aggregate (MTA) as direct pulp capping in young permanent teeth. J Clin Pediatr Dent. 2006 Winter;31(2):72-6. doi: 10.17796/jcpd.31.2.n462281458372u64. PMID 17315797
- [Background] Gruythuysen RJ, van Strijp AJ, Wu MK. Long-term survival of indirect pulp treatment performed in primary and permanent teeth with clinically diagnosed deep carious lesions. J Endod. 2010 Sep;36(9):1490-3. doi: 10.1016/j.joen.2010.06.006. PMID 20728715
- [Background] Lygidakis NA, Wong F, Jalevik B, Vierrou AM, Alaluusua S, Espelid I. Best Clinical Practice Guidance for clinicians dealing with children presenting with Molar-Incisor-Hypomineralisation (MIH): An EAPD Policy Document. Eur Arch Paediatr Dent. 2010 Apr;11(2):75-81. doi: 10.1007/BF03262716. PMID 20403301
- [Background] Mejare I, Cvek M. Partial pulpotomy in young permanent teeth with deep carious lesions. Endod Dent Traumatol. 1993 Dec;9(6):238-42. doi: 10.1111/j.1600-9657.1993.tb00279.x. PMID 8143574
- [Background] Nosrat A, Seifi A, Asgary S. Pulpotomy in caries-exposed immature permanent molars using calcium-enriched mixture cement or mineral trioxide aggregate: a randomized clinical trial. Int J Paediatr Dent. 2013 Jan;23(1):56-63. doi: 10.1111/j.1365-263X.2012.01224.x. Epub 2012 Feb 6. PMID 22309243
- [Background] Orstavik D, Kerekes K, Eriksen HM. The periapical index: a scoring system for radiographic assessment of apical periodontitis. Endod Dent Traumatol. 1986 Feb;2(1):20-34. doi: 10.1111/j.1600-9657.1986.tb00119.x. No abstract available. PMID 3457698
- [Background] Rajasekharan S, Martens LC, Cauwels RG, Verbeeck RM. Biodentine material characteristics and clinical applications: a review of the literature. Eur Arch Paediatr Dent. 2014 Jun;15(3):147-58. doi: 10.1007/s40368-014-0114-3. Epub 2014 Mar 11. PMID 24615290
- [Background] Rodd HD, Boissonade FM, Day PF. Pulpal status of hypomineralized permanent molars. Pediatr Dent. 2007 Nov-Dec;29(6):514-20. PMID 18254423
- [Background] Seow WK. Developmental defects of enamel and dentine: challenges for basic science research and clinical management. Aust Dent J. 2014 Jun;59 Suppl 1:143-54. doi: 10.1111/adj.12104. Epub 2013 Oct 27. PMID 24164394
- [Background] Sjogren U, Hagglund B, Sundqvist G, Wing K. Factors affecting the long-term results of endodontic treatment. J Endod. 1990 Oct;16(10):498-504. doi: 10.1016/S0099-2399(07)80180-4. PMID 2084204
- [Background] Taha NA, Ahmad MB, Ghanim A. Assessment of Mineral Trioxide Aggregate pulpotomy in mature permanent teeth with carious exposures. Int Endod J. 2017 Feb;50(2):117-125. doi: 10.1111/iej.12605. Epub 2016 Jan 30. PMID 26715408
- [Background] Ward J. Vital pulp therapy in cariously exposed permanent teeth and its limitations. Aust Endod J. 2002 Apr;28(1):29-37. doi: 10.1111/j.1747-4477.2002.tb00364.x. PMID 12360679
- [Background] Weerheijm KL, Duggal M, Mejare I, Papagiannoulis L, Koch G, Martens LC, Hallonsten AL. Judgement criteria for molar incisor hypomineralisation (MIH) in epidemiologic studies: a summary of the European meeting on MIH held in Athens, 2003. Eur J Paediatr Dent. 2003 Sep;4(3):110-3. PMID 14529329
- [Background] Weerheijm KL, Jalevik B, Alaluusua S. Molar-incisor hypomineralisation. Caries Res. 2001 Sep-Oct;35(5):390-1. doi: 10.1159/000047479. No abstract available. PMID 11641576
- [Background] William V, Messer LB, Burrow MF. Molar incisor hypomineralization: review and recommendations for clinical management. Pediatr Dent. 2006 May-Jun;28(3):224-32. PMID 16805354
- [Background] Witherspoon DE. Vital pulp therapy with new materials: new directions and treatment perspectives--permanent teeth. J Endod. 2008 Jul;34(7 Suppl):S25-8. doi: 10.1016/j.joen.2008.02.030. PMID 18565368